CLINICAL TRIAL: NCT04158674
Title: Interest of Levosimendan in Reducing Weaning Failures of ExtraCorporeal Life Support - ECLS. Randomized, Controlled, Multicenter, Double-blind, Multicenter Clinical Trial
Brief Title: Interest of Levosimendan in Reducing Weaning Failures of ExtraCorporeal Life Support - ECLS
Acronym: Weanilevo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: There was insufficient funding to continue the study in good conditions.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELLOUZE_ORION_2018
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan (Experimental)
  Interventions: Drug: Levosimendan
- Placebo (Sham Comparator)
  Interventions: Drug: Cernevit

INTERVENTIONS:
Drug: Levosimendan — Levosimendan 2.5mg/ml, solution to be diluted for infusion Dilution in a 500ml bag of 5% Glucose The product is administered as a continuous infusion for 24 hours at an initial rate of 0.2 µg/kg/min
  Arms: Levosimendan
Drug: Cernevit — mixture of 12 vitamins The dilution of the treatment is done in a 500ml bag of 5% Glucose The product is administered as a continuous infusion for 24 hours at an initial rate of 0.2 µg/kg/min
  Arms: Placebo

SUMMARY:
Extracorporeal life support (ECLS) is a circulatory cardio supplementation technique; it therefore makes it possible to compensate for a defective cardiac or cardio-respiratory function. ECLS nevertheless remains a temporary assistance technique pending a potential recovery of cardiac function, or it can be used to direct patients towards a heart transplant or long-term circulatory assistance (Left Ventricular Assist Device (LVAD) or Total Heart). In patients with complete or partial recovery of cardiac and circulatory function, ECLS withdrawal may be considered. Withdrawal from ECLS remains a delicate phase and the risk of failure is high. The mechanism of action of levosimendan, a drug that increases the contractility of the heart, suggests that it would improve the heart-vessel connection and reduce the rate of ECLS withdrawal failure. The effect of levosimendan is maximal 24 to 48 hours after the end of the infusion and has a prolonged period of action.

The objective is to evaluate the efficacy of levosimendan administration (0.2 µg/kg/min over 24 hours) - versus placebo - prior to ECLS removal on the rate of withdrawal failure in patients under ECLS.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* patient or person responsible for the patient has given written consent
* patient with acute circulatory heart failure under ECLS
* patient meeting criteria for ECLS withdrawal

  * ECLS flow rate at 1.0-1.5l/min and/or ECLS pump rpm ≤ 1500 rpm
  * LVEF > 20% in cardiac ultrasound and aortic ITV > 10 cm
  * VIS score ≤ 10
  * Arterial lactates ≤ 2 mmol/l
  * Right ventricular outflow tract shortening fraction > 30%
  * Basal diameter at the tricuspid telediastolic ring of the right ventricle < 35 mm
  * Fraction of inspired oxygen combined between ventilator and ECLS < 80%
* ECLS withdrawl scheduled within 48 hours
* Absence of an initial or progressive infectious episode (no planned introduction of antibiotic therapy within 48 hours prior to inclusion)

Exclusion Criteria:

* Patient with hepatic insufficiency: cytolysis at least 20 times normal
* Drug intoxication and attempted suicide
* Patient with a contraindication to the use of levosimendan:

  * hypersensitivity to the active substance or any of the excipients
  * severe hypotension and ventricular tachycardia
  * significant mechanical obstructions affecting ventricular filling and/or ejection
  * severe renal failure (creatinine clearance < 30 ml/min)
  * severe liver failure (TP<50%)
  * history of torsades de pointes
* Patient with a contraindication to the use of CERNEVIT®:

  * hypersensitivity to active substances, in particular to vitamin B1 or to one of the excipients or to soy protein products or to peanut protein products
  * hypervitaminosis to any vitamin contained in this formulation
  * severe hypercalcemia, hyper calciuria, tumour, bone metastasis, primary hyperparathyroidism, granulomatosis
* patient not affiliated to or not benefiting from national health insurance
* patient subject to legal protection (curatorship, guardianship)
* patient subject to limited judicial protection
* pregnant, parturient or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
ECLS withdrawal failure | 7 days after ECLS removal
  Withdrawal failure is defined as the absence of ECLS discontinuation within 48 hours of randomization or the use of temporary circulatory assistance such as ECLS, Impella® pump or intra-aortic balloon pump (IABP) or death

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Ellouze O, Soudry Faure A, Radhouani M, Abou-Arab O, Besnier E, Moussa M, Cransac A, Ksiazek E, Fischer MO, Mertes PM, Bouhemad B, Guinot PG. Levosimendan in venoarterial ECMO weaning. Rational and design of a randomized double blind multicentre trial. ESC Heart Fail. 2021 Aug;8(4):3339-3347. doi: 10.1002/ehf2.13427. Epub 2021 Jun 18. PMID 34145993